CLINICAL TRIAL: NCT07167446
Title: Exploring the Neuroprotective Potential of Cannabidiol (CBD) in Preventing Oxaliplatin (Ox)-Induced Neuropathy: A Prospective Study
Brief Title: Neuroprotective Potential of Cannabidiol (CBD) in Preventing Oxaliplatin (Ox)-Induced Neuropathy
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GI-249; 1R21CA292276-01A1 (NIH)
Record Dates: First submitted 2025-08-27; First posted 2025-09-11 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Oxaliplatin Induced Peripheral Neuropathy in Cancer Patients; Metastatic Colorectal Cancer (CRC); Peripheral Neuropathy Due to Chemotherapy
Keywords: Oxaliplatin-Induced Peripheral Neuropathy (OIPN); Cannabidiol (CBD); Colorectal Cancer (CRC); Neuroprotection
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (CBD) (Experimental): Participants receive hemp-derived cannabidiol (CBD) capsules in addition to standard oxaliplatin-based chemotherapy.
  Interventions: Drug: Cannabidiol (CBD); Drug: oxaliplatin-based chemotherapy
- Standard of Care (Active Comparator): Participants receive standard oxaliplatin-based chemotherapy without CBD supplementation
  Interventions: Drug: oxaliplatin-based chemotherapy

INTERVENTIONS:
Drug: Cannabidiol (CBD) — Oral hemp-derived CBD capsules, 150 mg twice daily (with titration in Cycle 1; dose reductions permitted for tolerability). Administered starting the day before oxaliplatin infusion and continued for 7 days after each chemotherapy cycle.
  Other Names: hemp-derived cannabidiol; CBD capsules
  Arms: Cannabidiol (CBD)
Drug: oxaliplatin-based chemotherapy — Standard of care oxaliplatin-based regimens per NCCN guidelines (e.g., FOLFOX or CAPEOX), administered in 2-3 week cycles for a maximum of 6 months.

SUMMARY:
This is a pilot, prospective, randomized study evaluating the feasibility and acceptability of incorporating hemp-derived cannabidiol (CBD) supplementation to prevent oxaliplatin-induced peripheral neuropathy (OIPN) in patients receiving oxaliplatin-based chemotherapy for colorectal cancer (CRC). Participants will be randomized to receive either CBD capsules in addition to standard therapy or standard therapy alone.

DETAILED DESCRIPTION:
Patients with metastatic colorectal cancer (mCRC) scheduled to receive at least 3 months of oxaliplatin-based chemotherapy will be enrolled on this prospective, randomized, open-label pilot study. A total of 30 patients will be randomized 2:1, with 20 patients assigned to the CBD supplementation arm and 10 patients assigned to the standard of care arm. Patients with pre-existing neuropathy, prior oxaliplatin exposure, or active cannabinoid use will be excluded.

Patients in the intervention arm will receive hemp-derived CBD capsules at a dose of 150 mg orally twice daily (following a titration during Cycle 1) starting the day before oxaliplatin and continuing through 7 days after each chemotherapy cycle. Standard oxaliplatin-based chemotherapy will be administered every 2-3 weeks per NCCN guidelines. Compliance will be monitored through pill counts, patient reporting, and scheduled check-ins. Dose adjustments to 100 mg or 50 mg twice daily will be permitted for treatment-related adverse events at investigator discretion.

Neuropathy will be assessed using both physician grading (CTCAE v5) and patient-reported outcomes (FACT-GOG NTx-13). Safety monitoring will include laboratory tests, neurological and physical examinations, and psychiatric evaluation with the Columbia Suicide Severity Rating Scale (C-SSRS). Exploratory analyses will measure circulating inflammatory cytokines (IL-6, TNF-α) and neuropathy-associated microRNAs (miR-155, miR-146a).

A total of 30 patients (20 intervention, 10 control) will be enrolled at Fox Chase Cancer Center over a 2-year period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with metastatic, locally advanced unresectable colorectal cancer patients planned to receive Ox based chemotherapy in metastatic setting (at least 3 months planned).
2. Subjects are allowed to have one cycle of Ox based chemotherapy before enrollment.
3. ECOG PS 0-2
4. No prior platinum exposure
5. No evidence of ongoing neuropathy of any grade at the time of enrollment
6. Patients must have marrow and organ function appropriate for systemic therapy, as per physician's discretion, but liver function should meet criteria below:

   1. Total Bilirubin: less than and/or equal to 1.5 X ULN
   2. AST(SGOT)/ALT(SGPT): less than and/or equal to 3 X ULN (5 X ULN in patients with liver metastases
7. Ability to understand and willingness to sign a written informed consent and HIPAA consent document.

   Exclusion Criteria:
8. Family history of genetic/familial neuropathy and personal history of ongoing neuropathy (any grade) or nervous system disease with the potential to affect cognition, Parkinson's disease, or multiple sclerosis.
9. Routine use of recreational marijuana products (deﬁned as > 4 times per month) or illicit drug use per self-reported history within the last 90 days. If using medical cannabis products, it should be stopped at least 1 week prior to inclusion.
10. Known underlying liver disease (Child-Pugh B or C) or baseline elevation of total bilirubin greater than and/or equal to 1.5 x upper limit of normal based on screening laboratory values.
11. 1Untreated brain metastases (can increase seizure risk), or treated brain metastases on anti-seizure medications.
12. Patients being treated with anti-seizure or anti-psychotic medications. Patients with a prior history of anti-seizure medication use, who have been off treatment for more than 3 months, are eligible. Use of Selective Serotonin Reuptake Inhibitors (SSRIs) is permitted.
13. Concomitant treatment with strong inducers of CYP3A4 and/or strong inducers of CYP2C19.
14. Underlying history of epilepsy/recurrent seizure disorder or unexplained seizure within past 6 months.
15. Patients with current or lifetime diagnosis of schizophrenia spectrum disorder, psychotic disorder, bipolar disorder type I & II, cluster B personality disorders (antisocial, borderline, narcissistic, histrionic), eating disorders, as defined by Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revised (DSM-5-TR, APA 2022)
16. Recent history or clinical concern for major depression with suicidal ideation as determined by investigator assessment at baseline
17. Currently taking medications known to be contraindicated with Epidiolex -FDA-approved CBD (buprenorphine, leflunomide, levomethadyl acetate, lomitapide, mipomersen, pexidartinib, propoxyphene, sodium oxybate, teriflunomide, clobazam, lamotrigine, valproate).
18. Women who are pregnant or breastfeeding, and individuals of any sex who are capable of reproduction and unwilling to use an effective form of birth control (e.g., condoms, diaphragm, birth control pills, or IUD).
19. Patients may not be receiving any other investigational agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2027-09-05 (Estimated); Study Completion 2028-09-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants adherent to the CBD supplementation protocol at Week 12, as determined by pill counts, patient self-report, and clinic compliance logs. | Baseline through Week 12 of treatment
Acceptability of CBD supplementation as measured by the Feasibility of Intervention Measure (FIM) | Baseline through Week 12 of treatment
  5-point Likert scale, each item is scored 1-5. Higher scores = higher acceptability and feasibility of implementing the intervention

SECONDARY OUTCOMES:
Incidence of physician-reported chemotherapy-induced peripheral neuropathy (CIPN), defined as Grade ≥2 by CTCAE v5.0. | From baseline through end of oxaliplatin-based chemotherapy and up to 4 weeks after treatment completion (short-term follow-up)
Change from baseline in patient-reported neuropathy symptoms using the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group Neurotoxicity (FACT-GOG NTx-13) scale | From baseline through end of oxaliplatin-based chemotherapy and up to 4 weeks after treatment completion (short-term follow-up)
  Each item is scored on a 5-point Likert scale (0 = Not at all to 4 = Very much).
  Total scores range from 0 to 52, with higher scores indicating more severe neuropathy symptoms
Incidence and profile of treatment-emergent adverse events (TEAEs), as classified by CTCAE v5.0 | From baseline through end of oxaliplatin-based chemotherapy and up to 4 weeks after treatment completion (short-term follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Namrata Vijayvergia, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States